CLINICAL TRIAL: NCT03498950
Title: Changes in Sense of Taste of Patients Submitted to Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fernanda de Paula Eduardo (Other)
Responsible Party: Sponsor-Investigator, Fernanda de Paula Eduardo, Dentist, Hospital Israelita Albert Einstein
Organization: Hospital Israelita Albert Einstein (Other)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 2591-16
Record Dates: First submitted 2018-04-02; First posted 2018-04-17 (Actual); Last update posted 2021-05-12 (Actual); Status verified 2021-05

CONDITIONS: Taste Disorders
MeSH Terms: conditions — Taste Disorders | interventions — Laser Therapy

STUDY DESIGN:
Intervention Model Description: The study sample will be composed of 80 patients selected at the Hematopoietic Stem Cell Transplantation Center of the "Hospital Israelita Albert Einstein". The patients will be randomized and distributed into two groups.
Who Masked: Participant
Masking Description: The patients will be randomized and distributed into two groups: Placebo Group (n=40) - submitted to the routine laser therapy protocol in addition to simulated laser irradiation on the taste papillae; Test Group (n= 40) - submitted to the same laser therapy protocol as that of the Placebo Group, however, laser irradiation on the taste papillae will be effective.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Group (No Intervention): submitted to the routine laser therapy protocol in addition to simulated laser irradiation on the taste papillae
- Test Group (Experimental): submitted to the same laser therapy protocol as that of the Placebo Group, however, laser irradiation on the taste papillae will be effective.
  Interventions: Other: laser therapy

INTERVENTIONS:
Other: laser therapy — laser irradiation on the taste papillae
  Arms: Test Group

SUMMARY:
During conditioning with chemotherapy and radiotherapy for the transplantation of hematopoietic stem cells (HSCT), oral changes, such as mucositis, xerostomia infections and dysgeusia may occur. Low level laser therapy is used to minimize the intensity of the lesions, prevent ulcerations in the mucosa, and diminish the time of healing. To verify the efficacy of low level laser therapy in the prevention of dysgeusia in patients undergoing allogenic HSCT and detect the frequency of dysgeusia, the flavors most changed, and the association of these changes with the clinical conditions of the patient. The study sample will be composed of 80 patients selected at the Hematopoietic Stem Cell Transplantation Center of the "Hospital Israelita Albert Einstein". The patients will be randomized and distributed into two groups: Placebo Group (n=40) - submitted to the routine laser therapy protocol in addition to simulated laser irradiation on the taste papillae; Test Group (n= 40) - submitted to the same laser therapy protocol as that of the Placebo Group, however, laser irradiation on the taste papillae will be effective. Daily intraoral exam will be performed in all the patients to evaluate mucositis, xerostomia and depapillation. The taste acuity test will determine the function of taste, using samples with the four basic flavors. This will be performed on the first day of conditioning (T0), during the stage of neutropenia (T1), at the time of discharge after transplantation (T2) and 100 days after transplantation (T3). A questionnaire will also be applied to evaluate the impact of changes in taste, smell and xerostomia on the quality of life. Our hypothesis is that the laser irradiation on the lingual papillae would help to prevent the changes in the cells of the taste papillae, preserving their morphology and function, which may attenuate the change in sense of taste and have a positive impact on the quality of life of patients during transplantation.

DETAILED DESCRIPTION:
uring conditioning with chemotherapy and radiotherapy for the transplantation of hematopoietic stem cells (HSCT), oral changes, such as mucositis, xerostomia infections and dysgeusia may occur. Low level laser therapy is used to minimize the intensity of the lesions, prevent ulcerations in the mucosa, and diminish the time of healing. To verify the efficacy of low level laser therapy in the prevention of dysgeusia in patients undergoing allogenic HSCT and detect the frequency of dysgeusia, the flavors most changed, and the association of these changes with the clinical conditions of the patient. The study sample will be composed of 80 patients selected at the Hematopoietic Stem Cell Transplantation Center of the "Hospital Israelita Albert Einstein". The patients will be randomized and distributed into two groups: Placebo Group (n=40) - submitted to the routine laser therapy protocol in addition to simulated laser irradiation on the taste papillae; Test Group (n= 40) - submitted to the same laser therapy protocol as that of the Placebo Group, however, laser irradiation on the taste papillae will be effective. Daily intraoral exam will be performed in all the patients to evaluate mucositis, xerostomia and depapillation. The taste acuity test will determine the function of taste, using samples with the four basic flavors. This will be performed on the first day of conditioning (T0), during the stage of neutropenia (T1), at the time of discharge after transplantation (T2) and 100 days after transplantation (T3). A questionnaire will also be applied to evaluate the impact of changes in taste, smell and xerostomia on the quality of life. Our hypothesis is that the laser irradiation on the lingual papillae would help to prevent the changes in the cells of the taste papillae, preserving their morphology and function, which may attenuate the change in sense of taste and have a positive impact on the quality of life of patients during transplantation.

ELIGIBILITY:
Inclusion Criteria:

* submitted a bone marrow transplantation
* adequate oral hygiene
* absence of periodontal disease and other infectious foci prior to transplantation
* normal chewing, swallowing and phonation functions prior to transplantation
* participation of all previously planned laser therapy sessions.

Exclusion Criteria:

* not performing all the steps of oral hygiene oriented during the transplant
* lack of collaboration in diagnostic test of the palate
* lack of records on dietary intake
* absence of record of clinical data of interest for the project in the medical record
* death during the transplant or 30 days after the completion of the bone marrow transplantation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
descriptive function of taste | 100 days
  using samples with the four basic flavors

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda de P Eduardo, Principal Investigator — Hospital Israelita Albert Einstein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epstein JB, Barasch A. Taste disorders in cancer patients: pathogenesis, and approach to assessment and management. Oral Oncol. 2010 Feb;46(2):77-81. doi: 10.1016/j.oraloncology.2009.11.008. Epub 2009 Dec 28. PMID 20036797
- [Background] Boer CC, Correa ME, Miranda EC, de Souza CA. Taste disorders and oral evaluation in patients undergoing allogeneic hematopoietic SCT. Bone Marrow Transplant. 2010 Apr;45(4):705-11. doi: 10.1038/bmt.2009.237. Epub 2009 Sep 21. PMID 19767788
- [Background] Just T, Pau HW, Bombor I, Guthoff RF, Fietkau R, Hummel T. Confocal microscopy of the peripheral gustatory system: comparison between healthy subjects and patients suffering from taste disorders during radiochemotherapy. Laryngoscope. 2005 Dec;115(12):2178-82. doi: 10.1097/01.MLG.0000181502.07160.86. PMID 16369163
- [Background] Schubert MM, Eduardo FP, Guthrie KA, Franquin JC, Bensadoun RJ, Migliorati CA, Lloid CM, Eduardo CP, Walter NF, Marques MM, Hamdi M. A phase III randomized double-blind placebo-controlled clinical trial to determine the efficacy of low level laser therapy for the prevention of oral mucositis in patients undergoing hematopoietic cell transplantation. Support Care Cancer. 2007 Oct;15(10):1145-54. doi: 10.1007/s00520-007-0238-7. Epub 2007 Mar 29. PMID 17393191